CLINICAL TRIAL: NCT03553264
Title: Impact of Home-based Three-dimensional Virtual Reality Procedures in Vestibular Rehabilitation Protocols: a Controlled Trial
Brief Title: Three-dimensional Virtual Reality Procedures in Vestibular Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uniter Onlus (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniterHMD
Record Dates: First submitted 2018-05-16; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Vestibular Diseases; Virtual Rehabilitation
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head Mounted Device (Experimental): In addition to the Vestibular Rehabilitation protocol, each HMD group patient will perform Virtual Reality Rehabilitation by means of the game protocol "Track Speed Racing 3D" uninterruptedly for 20min/day, while sitting on a chair or sofa, after the smartphone accommodation into the HMD 'Revelation' 3D VR Headset. The game consists of a point-of-view race in which the car is steered from the cockpit by tilting the head to the left and to the right to avoid swerving off the road and to achieve all the goals before finishing the lap. During this real car experience, the visual background and the scenario change perspective according to the patients' left or right tilted head movements, possibly emulating eye-head exercises that induce visual-vestibular conflicts.
  Interventions: Device: Virtual Reality Rehabilitation; Other: Vestibular Rehabilitation
- Vestibular Rehabilitation (Active Comparator): Patients will be actively involved in adapting the exercise program to suit their symptoms, capabilities, and lifestyle. Following previous protocols, the home exercise program will include a patient-tailored combination of adaptation (without and with the target moving in pitch and yaw planes for 1min each three times per day), substitution, habituation, and balance exercises, and all chronic unilateral vestibular hypofunction patients will be seen twice a week for 4 weeks for 30-45 min and monitored for adherence. Between supervised sessions, patients will perform a twice-daily home exercise program for a total of 30-40min/day.
  Interventions: Other: Vestibular Rehabilitation

INTERVENTIONS:
Device: Virtual Reality Rehabilitation — Track Speed Racing 3D game will run with HMD 'Revelation' 3D VR Headset and each HMD group patient will be instructed to perform the game protocol uninterruptedly for 20min/day, while sitting on a chair or sofa.
  Arms: Head Mounted Device
Other: Vestibular Rehabilitation — The home exercise program will include a patient-tailored combination of adaptation (without and with the target moving in pitch and yaw planes for 1min each three times per day), substitution, habituation, and balance exercises

SUMMARY:
The aim of the present study will be to discover possible (i) improvements achievable in unilateral vestibular hypofunction patients using a self-assessed head-mounted device (HMD)-based gaming procedure when combined with a classical vestibular rehabilitation protocol (HMD group) as compared with a group undergoing only vestibular rehabilitation and (ii) HMD procedure-related side effects. Main outcomes will be: otoneurological testing (vestibulo-ocular reflex gain study by means of vHIT and posturography measures with particular attention on power spectra) and self-report and performance measures (DHI, DGI and ABC). Side effects of HMD implementation will be studied by means of Simulator Sickness Questionnaires.

Moreover, second part of the study would collect patients' data one year after the end of the vestibular rehabilitation or its implementation with HMD.

DETAILED DESCRIPTION:
Due to the recent outbreak of virtual reality in the field of rehabilitation, the use of head-mounted devices has been proposed in addition to conventional vestibular rehabilitation therapy in unilateral vestibular hypofunction patients. This approach has been proved to be useful in maximizing vestibular rehabilitation outcomes, with minimum simulator-related side effects. Virtual reality-based devices have been tested in vestibular rehabilitation by many clinicians, due to the possibility of achieving habituation, substitution and adaptation, the effectiveness in people presenting visual vertigo, and the positive effects on anxiety.

Thus, due to the undeniable relevance of testing outcomes of vestibular rehabilitation, and the promising results of head-mounted device-based home exercises in ameliorating its effects, the aim of this study will be to compare - in terms of short- (one week) and long-term (one year) effects - the subjective and objective indicators of vestibular function in a population of patients with unilateral vestibular hypofunction after completing conventional vestibular rehabilitation therapy with a randomized group who underwent a mixed-methods protocol including vestibular rehabilitation and head-mounted device treatment over the same period of time.

ELIGIBILITY:
Inclusion Criteria:

- right-handed patients affected by right chronic Unilateral Vestibular Hypofunction, the diagnosis of which will be achieved with at least 25% reduced vestibular response at bithermal water caloric irrigations on one side when calculated by means of Jongkees' formula after at least 3 months from the onset of symptoms.

Exclusion Criteria:

* negative anamnesis for malignancy,
* negative anamnesis for head trauma,
* negative anamnesis for neuropsychiatric disorders
* negative anamnesis for metabolic diseases
* negative anamnesis for cardiovascular diseases
* negative anamnesis for endocrine diseases
* treatment with drugs possibly impacting on auditory and visuo-vestibular functions
* negative anamnesis for infectious diseases
* negative anamnesis for otoneurological diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Otoneurological Test | one month
  Study of vestibulo-ocular reflex VOR) by means of vHIT measuring its gain as the ratio between head and eye velocity. Low VOR gain values (range: 0.8-1) indicate low levels of activity of the semicircular canal.

SECONDARY OUTCOMES:
Balance Test | one month
  Study of the surface of the ellipse of confidence (mm) by means of static posturography platform will be used to assess the sway of the posture. Low levels of outcomes indicate better performances. No specific reference ranges are given in literature.
Self-report dizziness handicap | one month
  The Italian Dizziness Handicap Inventory (DHI) wil be used to assess the self-report dizziness handicap. It consists of 25 questions designed to assess a patient's functional (nine questions), emotional (nine questions), and physical (seven questions) limitations; scores range from 0 to 100, with moderate and severe disability usually associated with scores above 30 and 60, respectively
Balance Confidence | one month
  The Activities-specific Balance Confidence scale will be used to record the patient's perceived level of balance confidence during 16 everyday activities ranging from 0 to 100%. Higher values are referred to better balance confidence. No cut-off are given in literature.
Gait | one month
  The Dynamic Gait Index will examin the patient's ability to perform various gait activities on an eight-item scale; range is from 0 to 24, with scores less than 19 indicating increased risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Micarelli, M.D.,Ph.D., Principal Investigator — Uniter Onlus
Locations (1):
- UNITER ONLUS for balance and rehabilitation research, Guidonia, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergeron M, Lortie CL, Guitton MJ. Use of Virtual Reality Tools for Vestibular Disorders Rehabilitation: A Comprehensive Analysis. Adv Med. 2015;2015:916735. doi: 10.1155/2015/916735. Epub 2015 Apr 30. PMID 26556560
- [Result] Alahmari KA, Sparto PJ, Marchetti GF, Redfern MS, Furman JM, Whitney SL. Comparison of virtual reality based therapy with customized vestibular physical therapy for the treatment of vestibular disorders. IEEE Trans Neural Syst Rehabil Eng. 2014 Mar;22(2):389-99. doi: 10.1109/TNSRE.2013.2294904. PMID 24608691